CLINICAL TRIAL: NCT03950830
Title: Phase II Study of Disulfiram and Cisplatin in Refractory TGCTs.
Brief Title: Disulfiram and Cisplatin in Refractory TGCTs.
Acronym: DISGCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Slovakia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCT-SK-006
Record Dates: First submitted 2019-05-12; First posted 2019-05-15 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Germ Cell Tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Disulfiram

STUDY DESIGN:
Intervention Model Description: Non-randomized, open-label, single center trial to assess efficacy (as measured by overall response rate of disulfiram and cisplatin in patients with multiple relapsed/refractory germ cell tumors (GCTs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Cisplatin 50mg/m2 day 1 and 2, every 3 weeks, Disulfiram 400mg daily, continuously
  Interventions: Drug: Disulfiram

INTERVENTIONS:
Drug: Disulfiram — Disulfiram 400mg daily, continuously
  Other Names: Antabus

SUMMARY:
Non-randomized, open-label, single center trial to assess efficacy (as measured by overall response rate (ORR) by RECIST 1.1 of disulfiram and cisplatin in patients with multiple relapsed/refractory germ cell tumors (GCTs).

DETAILED DESCRIPTION:
Germ-cell tumours (GCTs) are extraordinarily chemosensitive and resemble the clinical and biological characteristics of a model for the cure of cancer. Nonetheless, a small proportion of patients do not have a durable complete remission (CR) with initial chemotherapy. Only 20-40% of them will be cured with the use of platinum-containing standard-dose or high-dose salvage chemotherapy with autologous stem cell transplantation (ASCT). Patients who fail to be cured after second-line salvage therapy have an extremely poor prognosis and long term survival had been documented in <5%. Paclitaxel plus ifosfamide and cisplatin is considered as a standard salvage chemotherapy in relapsed good prognosis GCTs, however, up to 40% of favourable prognosis patients failed to achieve durable response to this combination, and therefore new treatment strategies are warranted.

Previously, it was showed that cisplatin resistant TGCTs overexpress ALDH isoforms and inhibition of ALDH activity by disulfiram is associated with reconstitution of cisplatin sensitivity. Cisplatin-resistant TGCTs exhibited increased sensitivity to ALDH inhibitor disulfiram in vitro. Although Disulfiram (Antabuse) is an approved drug to support the treatment of chronic alcoholism, it may serve as an antitumor agent suitable for the drug repurposing in combination therapy in order to inhibit ALDH activity thus overcoming a cisplatin resistance in refractory TGCTs. Indeed, disulfiram in combination with cisplatin very efficiently eradicated platinum-resistant NTERA-2 model spheroids and significantly inhibited xenograft growth in vivo in our experimental system.

Based on aforementioned data, investigators suggest that there is strong rationale to inhibit ALDH in TGCT. Investigators hypothesize that inactivation of ALDH by disulfiram recover cisplatin sensitivity in patients with progressing or relapsing germ cell cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent .
2. Men aged 18 years or older.
3. ECOG performance status: 0-1.
4. Histologically confirmed extracranial primary germ cell cancer, seminoma, or nonseminoma.
5. Rising serum markers (i.e., alpha-fetoprotein and human chorionic gonadotropin) on sequential measurement or biopsy-proven unresectable germ cell cancer.
6. Multiple relapsed/refractory GCTs (at least 2 lines of previous chemotherapy and/or patients relapsing after high-dose chemotherapy or for patients non fit enough for high-dose chemotherapy.
7. Primary mediastinal GCTs in first relapse.
8. Patient's disease must not be amenable to cure with either surgery or chemotherapy in the opinion of investigator.
9. RECIST 1.1 Measurable disease.
10. Adequate hematologic function defined by ANC > 1500/mm3, platelet count > 100 000/mm3 and hemoglobin level > 9g/dl.
11. Adequate liver function defined by a total bilirubin level < 1.5 ULN, and ALT, AST < 3 ULN or < 5 in case of liver metastases. For subjects with Gilbert's syndrome bilirubin > 1.5 × ULN is allowed if no symptoms of compromised liver function are present.
12. Adequate renal function: measured or calculated (by Cockcroft formula) creatinine clearance > 50 ml/min. Cockcroft formula: CLcr = [(140-age) x weight (Kg)]/[72 x creat (mg/dl)].
13. At least 4 weeks must have elapsed since the last radiotherapy and/or chemotherapy before study entry.
14. At least 4 weeks must have elapsed since the last major surgery.
15. Complete recovery from prior surgery, and/or reduction of all adverse events from previous systemic therapy or radiotherapy to grade 1.
16. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

1. Patients who do not fit inclusion criteria.
2. Addiction to alcohol or drugs.
3. Other prior malignancy except successfully treated nonmelanoma skin cancer .
4. Need for metronidazole, warfarin and/or theophylline medication, the metabolism of which is likely influenced by disulfiram.
5. Patients who are taking medications metabolized by cytochrome P450 2E1, including chlorzoxazone or halothane and its derivatives.
6. Other concurrent approved or investigational anticancer treatment, including surgery, radiotherapy, chemotherapy, biologic-response modifiers, hormone therapy, or immunotherapy.
7. Female patients.
8. Patients infected by the Human Immunodeficiency Virus (HIV).
9. Patients with other severe acute or chronic medical condition, or laboratory abnormality that would impair, in the judgment of investigator, excess risk associated with study treatment, or which, in judgment of the investigator, would make the patient inappropriate for entry into this study.
10. Inability of oral intake, or drug absorbtion (e.g. malabsorption syndrome).
11. Hypersensitivity to any compound of the drug.
12. Sexually active men not using highly effective birth control if their partners are women of child-bearing potential.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 24 months
  Overall response rate by RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival | 24 months
  Progression-free survival
Overall survival | 24 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mego, Prof, Principal Investigator — National Cancer Institute, Slovakia
Locations (1):
- National Cancer Institute, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No